CLINICAL TRIAL: NCT05812781
Title: A Phase 2A, Single-Arm Study to Evaluate the Safety and Clinical Activity of VTX2735 in Participants With Cryopyrin-Associated Periodic Syndrome (CAPS)
Brief Title: A Study to Evaluate VTX2735 in Patients With Cryopyrin-associated Periodic Syndrome
Acronym: Explore
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zomagen Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VTX2735-201
Record Dates: First submitted 2023-03-28; First posted 2023-04-14 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cryopyrin Associated Periodic Syndrome
Keywords: Cryopyrin-Associated Periodic Syndrome; Ventyx; Zomagen; VTX2735; CAPS
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: VTX2735
- Cohort 2 (Experimental)
  Interventions: Drug: VTX2735

INTERVENTIONS:
Drug: VTX2735 — Dose A
  Arms: Cohort 1
Drug: VTX2735 — Dose B
  Arms: Cohort 2

SUMMARY:
This is a study to understand if taking VTX2735 is safe and effective in participants diagnosed with Cryopyrin-Associated Period Syndrome (CAPS). Approximately 10 patients will take VTX2735 Dose A or VTX2735 Dose B.

The study consists of a screening/washout period of up to 28 weeks, a 2 week treatment period, a treatment withdrawal period of up to 2 weeks, another 2 week treatment period, and a 4 week follow up period. The maximum length of treatment is 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of CAPS and FCAS subtype and mild clinical phenotype
* At least one flare during screening/washout
* Women must not be of childbearing potential or must agree to use two methods of highly effective contraception during the study and for 30 days after the last dose of the study product
* Men with a partner who is of childbearing potential must agree to use condoms plus another highly effective form of birth control during the study and for 90 days after the last dose of study product

Exclusion Criteria:

* Unwilling to comply with washout of anti-IL-1 therapy and tolerate symptoms of disease flare
* Moderate or severe CAPS manifestations or significant damage or any CAPS feature that presents a contraindication to washout of anti-IL-1 therapy
* Has a history of chronic or recurrent infectious disease
* Has a known immune deficiency or is immunocompromised
* Has hepatitis B or hepatitis C infection, human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS), or active tuberculosis (TB)
* Has another clinically important medical disorder that would compromise safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-03-18 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of VTX2735 | From the initial administration of VTX2735 through study completion, up to 10 weeks
  Incidence and severity of treatment-emergent adverse events (TEAE), serious adverse events (SAE), and discontinuation due to adverse events

SECONDARY OUTCOMES:
Mean change in the mean key symptom score (KSS) derived from the Daily Health Assessment Form, Second Generation (DHAF2) from baseline | From Day 1 to completion of treatment with VTX2735, up to Day 28
  Assess the change from baseline in disease activity using DHAF2 and KSS.
Achievement of 30%, 50%, or 75% improvement in mean KSS from baseline | From Day 1 to completion of treatment with VTX2735, up to Day 28
  Proportion of patients achieving 30%, 50%, or 75% improvement from baseline in disease activity using DHAF2 and KSS.
Number of days when the daily KSS is >3 | From Day 1 to completion of treatment with VTX2735, up to Day 28
  Number of multi-system disease flare days as defined by KSS
Number of days when any single DHAF2 symptom score is >3 | From Day 1 to completion of treatment with VTX2735, up to Day 28
  Number of single system disease flare days as defined by KSS
Maximum severity of any symptom score on DHAF2 | From Day 1 to completion of treatment with VTX2735, up to Day 28
  Maximum single DHAF2 symptom score

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Sonnergren, MD, PhD, Study Director — Ventyx Biosciences, Inc
Locations (2):
- United States (2):
  - Local Site # 222, San Diego, California
  - Local Site # 223, Columbus, Georgia

IPD SHARING:
Plan to Share IPD: Undecided